CLINICAL TRIAL: NCT06545721
Title: The Effect and Mechanism Of Weight Cycling on Hyperandrogenemia And Insulin Resistance in Polycystic Ovary Syndrome
Brief Title: Weight Cycling on Hyperandrogenemia and Insulin Resistance in Polycystic Ovary Syndrome
Acronym: WHIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wei Chen, Professor, Peking Union Medical College Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K5204
Record Dates: First submitted 2024-07-22; First posted 2024-08-09 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Weight Cycling; Hyperandrogenemia; Insulin Resistance; High-protein diet; Transcriptome; Metabolome; Inflammatory status
MeSH Terms: conditions — Polycystic Ovary Syndrome; Weight Cycling; Insulin Resistance | interventions — Exercise; Behavior Therapy

STUDY DESIGN:
Intervention Model Description: the sample size for the normal weight group is 45, and the sample size for the overweight/obese group is 380.
Masking Description: ancillary randomized substudy nested in WHIP cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal weight group (Experimental): 18.5 kg/m2 ≤ BMI < 24 kg/m2
  Interventions: Other: Adjusting dietary structure + exercise + behavioral intervention
- Obese/Overweight Group (Experimental): BMI ≥24 kg/m²
  Interventions: Other: Adjusting dietary structure + exercise + behavioral intervention
- Precision dietary prescription (nested substudy) (Experimental): Within the WHIP cohort, participants with PCOS and insulin resistance who enroll in the ancillary 12-week pragmatic intervention will receive a precision dietary prescription tailored to their baseline insulin-resistance metabolic subphenotype. The prescription includes an individualized daily energy deficit according to the Chinese guideline for medical nutrition therapy in overweight/obesity, personalized macronutrient distribution, and food-based meal plans. Participants receive dietitian counseling at baseline and scheduled follow-ups throughout the 12-week period, in addition to standard lifestyle advice provided in the parent cohort.
  Interventions: Behavioral: Precision dietary prescription
- Standard guideline-based low-energy diet (nested substudy control) (Active Comparator): Within the WHIP cohort, participants with PCOS and insulin resistance who enroll in the ancillary 12-week pragmatic intervention will receive a uniform low-energy diet based on standard guideline recommendations. The daily energy deficit is set according to the Chinese guideline for medical nutrition therapy in overweight/obesity, without tailoring to metabolic subphenotype. Contact frequency and follow-up intensity are comparable to the precision-diet arm, and standard lifestyle advice is provided throughout the 12-week period.
  Interventions: Behavioral: Standard guideline-based low-energy diet

INTERVENTIONS:
Other: Adjusting dietary structure + exercise + behavioral intervention — Adjusting to a healthy diet involves consuming low GI and low-fat foods, avoiding sugary drinks, increasing dietary fiber intake, reducing saturated fat while increasing omega-3 unsaturated fat intake, and limiting trans fat consumption. A weight loss program includes a high-protein diet, exercise, and behavioral intervention with daily total energy needs calculated based on ideal body weight (kg) x 15-20 kcal/kg/d; developing a daily meal plan with regular protein supplementation; limiting salt intake to ≤5 g/d; ensuring adequate water consumption at 2-3L/d; aiming for a dietary fiber intake of 25-30g/d; recommending micronutrient supplementation as needed; maintaining daily aerobic exercise (40 minutes at 70-80% HRmax) along with resistance training (20 minutes); establishing an early bedtime before 11pm and an early wake-up time.
  Arms: Normal weight group; Obese/Overweight Group
Behavioral: Precision dietary prescription — A 12-week precision diet program individualized to baseline insulin-resistance metabolic subphenotype, including personalized macronutrient targets, food-based meal plans, and dietitian-led counseling with regular follow-ups.
  Arms: Precision dietary prescription (nested substudy)
Behavioral: Standard guideline-based low-energy diet — A 12-week standardized low-energy diet based on national guideline recommendations for overweight/obesity, with the same counseling frequency as the precision-diet arm but without metabolic tailoring.
  Arms: Standard guideline-based low-energy diet (nested substudy control)

SUMMARY:
This study prospectively includes PCOS patients with normal weight and overweight/obesity, closely follows up and intensively manages them, and observes the level and distribution of weight reduction achieved by patients after lifestyle intervention (high-protein diet for weight loss). Additionally, it aims to provide reference for setting weight loss targets for future PCOS patients by comparing the differences in clinical improvement among patients achieving different degrees of weight reduction (<2% [equivalent to no weight loss], 2-5%, 5-10%, ≥10%) at different time points (3 months, 6 months) following dietary intervention. Furthermore, this study will compare the differences in reproductive and metabolic marker improvements between baseline PCOS patients experiencing weight rebound, those who successfully lost weight, and those who experienced weight rebound. This will help explore the impact of weight cycling on PCOS-related manifestations. Finally, at a genetic level, the study will analyze potential mechanisms underlying different outcome indicators by comparing differences in metagenomics, transcriptomics, and metabolomics among patient groups.

Ancillary/Nested Sub-study (12-week Precision Nutrition Trial):

Within the WHIP cohort, we will conduct a nested, prospective interventional sub-study to evaluate the efficacy of an insulin-resistance-phenotype-guided precision dietary prescription versus a standard guideline-based energy-restricted diet. Eligible participants are women with PCOS and insulin resistance enrolled in the cohort. The sub-study lasts 12 weeks with assessments at baseline and week 12. Primary endpoints include change in HOMA-IR and change in the core11 metabolic risk composite. Secondary endpoints include changes in gonadotropins (FSH, LH), sex steroid hormones (e.g., estradiol, progesterone), and patient-reported symptom scores.

DETAILED DESCRIPTION:
This study is a single-center, prospective cohort study that enrolled PCOS patients after screening. The patients were categorized into two groups based on their BMI: a normal weight group (18.5 kg/m2 ≤ BMI < 24 kg/m2) with a sample size of 45 and an overweight/obese group (BMI ≥ 24 kg/m2) with a sample size of 380, totaling 425 cases.

For the normal weight PCOS patients, interventions included control of total energy intake, adjustment of dietary structure, exercise, and behavioral intervention to prevent weight gain over a follow-up period of three months. If weight gain occurred during the follow-up period, these patients were transferred to the overweight/obese group for intensified intervention.

The overweight/obese PCOS patients received intensive intervention in accordance with high-protein diet adaptation criteria. This involved high-protein diets combined with exercise and behavioral intervention for weight reduction. After three months of follow-up, if they achieved their weight-loss goal, they transitioned to a low-energy diet and exercise intervention program to maintain their weight. If the goal was not met after three months, they continued with the high-protein weight-loss program.

The study compared differences in improvement in indicators such as insulin resistance (IR), blood androgen levels, inflammatory factors among different degrees of weight loss (<2%, 2% ≤weight loss <5%, 5%≤weight loss<10%, ≥10%), analyzing potential mechanisms.

For individuals experiencing weight cycling, differences in IR levels before and after rebounding from body mass were compared alongside changes in androgen levels and other metabolic indicators. This aimed to explore the impact of body mass cycling on clinical indicators while analyzing potential causes.

Ancillary/Nested Sub-study (12-week Precision Nutrition Trial):

A subset of cohort participants meeting criteria for PCOS with insulin resistance will enter a 12-week dietary intervention sub-study. Participants will be allocated in a 1:1 ratio to: (1) a phenotype-guided precision dietary prescription tailored to the individual's insulin-resistance metabolic subtype; or (2) a standard low-energy diet based on current Chinese clinical guidelines for overweight/obesity medical nutrition therapy. Both groups receive standardized lifestyle counseling and follow-up. Study visits occur at baseline and week 12. This nested sub-study is designed to test whether subtype-matched dietary prescriptions yield greater improvements in insulin resistance and metabolic risk than a uniform guideline diet, while remaining integrated within the parent WHIP cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-45 years in the reproductive period;
2. Women who have previously met the Rotterdam diagnostic criteria (at least 2 of the following 3 criteria have been confirmed, and have been diagnosed with PCOS): 1) Oligomenorrhea and/or anovulation; 2) clinical and/or biochemical evidence of hyperandrogenism; 3) ultrasound showing the presence of unilateral or bilateral polycystic ovaries;
3. Inclusion of 50 women in the normal weight group: 18.5 kg/m² ≤ BMI < 24 kg/m²; Inclusion of 400 women in the overweight/obese group: BMI ≥ 24 kg/m²;
4. Voluntarily participate in the intervention and sign an informed consent form.

Exclusion Criteria:

1. Currently pregnant or lactating, or have had a recent (within 6 months) plan for pregnancy;
2. Currently using known prescription weight loss medications (such as GLP-1RA, orlistat, topiramate, etc.);
3. History of weight loss surgery;
4. History of severe cardiovascular or cerebrovascular diseases; severe liver or kidney dysfunction (ALT > 3 times the upper limit of normal, or creatinine > 1.5 times the upper limit of normal); chronic or active gastrointestinal inflammatory diseases; severe systemic diseases; active malignant tumors;
5. Secondary obesity: including hypothalamic or pituitary obesity, obesity secondary to glucocorticoid use, hypogonadism-induced obesity, etc.;
6. Known history of serious endocrine system diseases;
7. Poor compliance with planned dietary interventions (psychiatric disorders such as binge eating disorder, anorexia nervosa, severe anxiety/depression);
8. Unable to follow up on time or deemed non-cooperative by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 425 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Weight loss rate | 6 month
  Percentage of weight loss: (Weight after reduction - Baseline weight before reduction) / Baseline weight before reduction (%)
Levels of insulin resistance | 6 month
  Measuring the level of insulin resistance in patients after the intervention.

SECONDARY OUTCOMES:
Fasting insulin level（FINS） | 6 month
  Measure the fasting insulin levels of patients after the intervention.
Fasting blood sugar（FBG） | 6 month
  Measure the fasting blood glucose level of the patient after the intervention.
Blood levels of androgen hormones (total testosterone, free testosterone index) | 6 month
  Measure the blood testosterone levels of the patients after the intervention.
Blood lipid levels (LDL-C, HDL-C, total cholesterol) | 6 month
  Measure lipid levels in patients after the intervention.
Levels of inflammatory factors (CRP, IL-6, TAC, GSH) | 6 month
  Detect the level of inflammatory factors in patients after intervention.
BMI | 6 month
  Measuring the BMI of patients after the intervention.
Waist | 6 month
  Measure the waist of the patients after the intervention.
waist-to-hip ratio | 6 month
  Measure the waist-to-hip ratio of the patients after the intervention.
Body fat percentage and distribution | 6 month
  Measure the Body Fat Content and Proportion in Patients after Intervention
Weight rebound rate | 6 month
  Determine the rate of weight rebound in patients after intervention. Weight rebound is defined as a rebound in weight (≥5kg or 5% above baseline weight) after weight loss.

OTHER OUTCOMES:
Change in insulin resistance (HOMA-IR) | 12 weeks
  Change from baseline to week 12 in HOMA-IR among participants enrolled in the ancillary precision-diet substudy.
Change in core metabolic risk profile | 12 weeks
  Change from baseline to week 12 in the composite Z-score of the 11 predefined metabolic indicators (BMI, waist, FINS, FPG, TG, HDL, LDL, ALT, SBP, UA, SHBG) in the ancillary substudy.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lizneva D, Suturina L, Walker W, Brakta S, Gavrilova-Jordan L, Azziz R. Criteria, prevalence, and phenotypes of polycystic ovary syndrome. Fertil Steril. 2016 Jul;106(1):6-15. doi: 10.1016/j.fertnstert.2016.05.003. Epub 2016 May 24. PMID 27233760
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS consensus workshop group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome (PCOS). Hum Reprod. 2004 Jan;19(1):41-7. doi: 10.1093/humrep/deh098. PMID 14688154
- [Background] Moran LJ, Misso ML, Wild RA, Norman RJ. Impaired glucose tolerance, type 2 diabetes and metabolic syndrome in polycystic ovary syndrome: a systematic review and meta-analysis. Hum Reprod Update. 2010 Jul-Aug;16(4):347-63. doi: 10.1093/humupd/dmq001. Epub 2010 Feb 16. PMID 20159883
- [Background] Barry JA, Kuczmierczyk AR, Hardiman PJ. Anxiety and depression in polycystic ovary syndrome: a systematic review and meta-analysis. Hum Reprod. 2011 Sep;26(9):2442-51. doi: 10.1093/humrep/der197. Epub 2011 Jul 1. PMID 21725075
- [Background] Teede HJ, Misso ML, Costello MF, Dokras A, Laven J, Moran L, Piltonen T, Norman RJ; International PCOS Network. Recommendations from the international evidence-based guideline for the assessment and management of polycystic ovary syndrome. Hum Reprod. 2018 Sep 1;33(9):1602-1618. doi: 10.1093/humrep/dey256. PMID 30052961
- [Background] Azziz R, Carmina E, Chen Z, Dunaif A, Laven JS, Legro RS, Lizneva D, Natterson-Horowtiz B, Teede HJ, Yildiz BO. Polycystic ovary syndrome. Nat Rev Dis Primers. 2016 Aug 11;2:16057. doi: 10.1038/nrdp.2016.57. PMID 27510637
- [Background] Randeva HS, Tan BK, Weickert MO, Lois K, Nestler JE, Sattar N, Lehnert H. Cardiometabolic aspects of the polycystic ovary syndrome. Endocr Rev. 2012 Oct;33(5):812-41. doi: 10.1210/er.2012-1003. Epub 2012 Jul 24. PMID 22829562
- [Background] Cowan S, Lim S, Alycia C, Pirotta S, Thomson R, Gibson-Helm M, Blackmore R, Naderpoor N, Bennett C, Ee C, Rao V, Mousa A, Alesi S, Moran L. Lifestyle management in polycystic ovary syndrome - beyond diet and physical activity. BMC Endocr Disord. 2023 Jan 16;23(1):14. doi: 10.1186/s12902-022-01208-y. PMID 36647089
- [Background] Stepto NK, Cassar S, Joham AE, Hutchison SK, Harrison CL, Goldstein RF, Teede HJ. Women with polycystic ovary syndrome have intrinsic insulin resistance on euglycaemic-hyperinsulaemic clamp. Hum Reprod. 2013 Mar;28(3):777-84. doi: 10.1093/humrep/des463. Epub 2013 Jan 12. PMID 23315061
- [Background] Teede HJ, Joham AE, Paul E, Moran LJ, Loxton D, Jolley D, Lombard C. Longitudinal weight gain in women identified with polycystic ovary syndrome: results of an observational study in young women. Obesity (Silver Spring). 2013 Aug;21(8):1526-32. doi: 10.1002/oby.20213. Epub 2013 Jul 2. PMID 23818329
- [Background] Lim SS, Davies MJ, Norman RJ, Moran LJ. Overweight, obesity and central obesity in women with polycystic ovary syndrome: a systematic review and meta-analysis. Hum Reprod Update. 2012 Nov-Dec;18(6):618-37. doi: 10.1093/humupd/dms030. Epub 2012 Jul 4. PMID 22767467
- [Background] Kazemi M, Hadi A, Pierson RA, Lujan ME, Zello GA, Chilibeck PD. Effects of Dietary Glycemic Index and Glycemic Load on Cardiometabolic and Reproductive Profiles in Women with Polycystic Ovary Syndrome: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Adv Nutr. 2021 Feb 1;12(1):161-178. doi: 10.1093/advances/nmaa092. PMID 32805007
- [Background] Lim SS, Hutchison SK, Van Ryswyk E, Norman RJ, Teede HJ, Moran LJ. Lifestyle changes in women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2019 Mar 28;3(3):CD007506. doi: 10.1002/14651858.CD007506.pub4. PMID 30921477
- [Background] Goss AM, Chandler-Laney PC, Ovalle F, Goree LL, Azziz R, Desmond RA, Wright Bates G, Gower BA. Effects of a eucaloric reduced-carbohydrate diet on body composition and fat distribution in women with PCOS. Metabolism. 2014 Oct;63(10):1257-64. doi: 10.1016/j.metabol.2014.07.007. Epub 2014 Jul 18. PMID 25125349
- [Background] Gokee-LaRose J, Gorin AA, Raynor HA, Laska MN, Jeffery RW, Levy RL, Wing RR. Are standard behavioral weight loss programs effective for young adults? Int J Obes (Lond). 2009 Dec;33(12):1374-80. doi: 10.1038/ijo.2009.185. PMID 19786967
- [Background] Robinson S, Chan SP, Spacey S, Anyaoku V, Johnston DG, Franks S. Postprandial thermogenesis is reduced in polycystic ovary syndrome and is associated with increased insulin resistance. Clin Endocrinol (Oxf). 1992 Jun;36(6):537-43. doi: 10.1111/j.1365-2265.1992.tb02262.x. PMID 1424179
- [Background] Moran LJ, Noakes M, Clifton PM, Wittert GA, Tomlinson L, Galletly C, Luscombe ND, Norman RJ. Ghrelin and measures of satiety are altered in polycystic ovary syndrome but not differentially affected by diet composition. J Clin Endocrinol Metab. 2004 Jul;89(7):3337-44. doi: 10.1210/jc.2003-031583. PMID 15240612
- [Background] Saarni SE, Rissanen A, Sarna S, Koskenvuo M, Kaprio J. Weight cycling of athletes and subsequent weight gain in middleage. Int J Obes (Lond). 2006 Nov;30(11):1639-44. doi: 10.1038/sj.ijo.0803325. Epub 2006 Mar 28. PMID 16568134
- [Background] Li W, Chen W. Weight cycling based on altered immune microenvironment as a result of metaflammation. Nutr Metab (Lond). 2023 Feb 22;20(1):13. doi: 10.1186/s12986-023-00731-6. PMID 36814270
- [Background] Matsuo T, Kato Y, Murotake Y, Kim MK, Unno H, Tanaka K. An increase in high-density lipoprotein cholesterol after weight loss intervention is associated with long-term maintenance of reduced visceral abdominal fat. Int J Obes (Lond). 2010 Dec;34(12):1742-51. doi: 10.1038/ijo.2010.95. Epub 2010 Jun 1. PMID 20514050
- [Background] El Ghoch M, Calugi S, Dalle Grave R. Weight cycling in adults with severe obesity: A longitudinal study. Nutr Diet. 2018 Jul;75(3):256-262. doi: 10.1111/1747-0080.12387. Epub 2017 Nov 8. PMID 29114979
- [Background] Kroeger CM, Hoddy KK, Varady KA. Impact of weight regain on metabolic disease risk: a review of human trials. J Obes. 2014;2014:614519. doi: 10.1155/2014/614519. Epub 2014 Aug 14. PMID 25197563
- [Background] Mehrabani HH, Salehpour S, Amiri Z, Farahani SJ, Meyer BJ, Tahbaz F. Beneficial effects of a high-protein, low-glycemic-load hypocaloric diet in overweight and obese women with polycystic ovary syndrome: a randomized controlled intervention study. J Am Coll Nutr. 2012 Apr;31(2):117-25. doi: 10.1080/07315724.2012.10720017. PMID 22855917
- [Background] Thomson RL, Buckley JD, Noakes M, Clifton PM, Norman RJ, Brinkworth GD. The effect of a hypocaloric diet with and without exercise training on body composition, cardiometabolic risk profile, and reproductive function in overweight and obese women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2008 Sep;93(9):3373-80. doi: 10.1210/jc.2008-0751. Epub 2008 Jun 26. PMID 18583464
- [Background] Makhija N, Tayade S, Toshniwal S, Tilva H. Clinico-Metabolic Profile in Lean Versus Obese Polycystic Ovarian Syndrome Women. Cureus. 2023 Apr 19;15(4):e37809. doi: 10.7759/cureus.37809. eCollection 2023 Apr. PMID 37214034
- [Result] Teede H, Deeks A, Moran L. Polycystic ovary syndrome: a complex condition with psychological, reproductive and metabolic manifestations that impacts on health across the lifespan. BMC Med. 2010 Jun 30;8:41. doi: 10.1186/1741-7015-8-41. PMID 20591140
- [Result] Pirotta S, Barillaro M, Brennan L, Grassi A, Jeanes YM, Joham AE, Kulkarni J, Couch LM, Lim SS, Moran LJ. Disordered Eating Behaviours and Eating Disorders in Women in Australia with and without Polycystic Ovary Syndrome: A Cross-Sectional Study. J Clin Med. 2019 Oct 14;8(10):1682. doi: 10.3390/jcm8101682. PMID 31615157